CLINICAL TRIAL: NCT01982786
Title: Randomized Phase II Feasibility Trial Of Image Guided External Beam Radiotherapy With Or Without High Dose Rate Brachytherapy Boost In Men With Intermediate-Risk Prostate Cancer
Brief Title: Feasibility Trial Of Image Guided External Beam Radiotherapy With Or Without High Dose Rate Brachytherapy Boost In Men With Intermediate-Risk Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR15
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): IGRT* 60 Gy in 20 fractions OR IGRT 78 Gy in 39 fractions
  Interventions: Radiation: Image guided external beam radiotherapy with or without brachytherapy boost
- Arm 2 (Active Comparator): IGRT 37.5 Gy in 15 fractions
  + HDR brachytherapy boost 15 Gy
  Interventions: Radiation: Image guided external beam radiotherapy with or without brachytherapy boost; Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Image guided external beam radiotherapy with or without brachytherapy boost — image guided external beam radiotherapy (IGRT) or IGRT with high dose rate (HDR) brachytherapy boost
Radiation: Brachytherapy — Brachytherapy boost
  Arms: Arm 2

SUMMARY:
This research is being done because investigators involved in this study would like to compare image guided external beam radiation therapy (IGRT) to IGRT plus HDR brachytherapy boost to see which treatment is better and what the side effects of treatment are.

DETAILED DESCRIPTION:
Before a big study is done, a smaller study (called a "feasibility study") is required to make sure that patients and physicians are willing to participate in a study comparing the two kinds of treatments, and to verify how the radiation therapy is given in different centres across Canada.

The standard or usual treatment for this disease includes treatment with IGRT or IGRT plus HDR brachytherapy boost.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma. The date of the last biopsy that verifies that the eligibility criterions have been met must be within 9 months prior to randomization. There must be no prior treatment.
* Intermediate-risk cancer patients based on the NCCN Guidelines (www.nccn.org):

  • TNM classification:
* T2b-T2c and Gleason Score < 8/10 and PSA < 20 ng/ml; or
* T1c-T2a and Gleason Score 7/10 and PSA < 20 ng/ml; or
* T1c-T2a and Gleason Score ≤ 6/10 and 10 ≤ PSA < 20 ng/ml

For patients who have been on alpha reductase inhibitors within the last 6 months, use the following guidelines:

* T2b-T2c and Gleason Score < 8/10 and PSA ≤ 10 ng/ml; or
* T1c-T2a and Gleason Score 7/10 and PSA ≤ 10 ng/ml; or
* T1c-T2a and Gleason Score ≤ 6/10 and 5 ≤ PSA ≤ 10 ng/ml
* No alpha reductase inhibitors (i.e. avodart, proscar) use within 2 weeks of randomization. A washout period of 2 weeks is required prior to randomization.
* Prostate volume ≤ 75 cc.
* American Urological Association (AUA) Symptom Index score < 20.
* Judged to be medically fit for IGRT and HDR brachytherapy boost by a radiation oncologist.
* ECOG Performance Status of 0 or 1.
* ≥ 18 years of age.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Protocol treatment is to begin within 4 weeks of patient randomization. HDR brachytherapy boost treatment is to begin within 3 weeks before or after IGRT for those randomized to Arm 2.
* Participants must be willing to take precautions to prevent pregnancy while on treatment. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention). However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures, he is responsible for beginning contraceptive measures.

Exclusion Criteria:

* History of transurethral resection of the prostate (TURP).
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Prior or current bleeding diathesis.
* Prior pelvic or prostate radiotherapy.
* Previous history of (or planned) androgen deprivation therapy.
* Evidence of metastatic disease.
* Any serious active disease or co-morbid medical condition, laboratory abnormality, psychiatric illness, active or uncontrolled infections, or serious illnesses or medical conditions that would prevent the patient from participating or to be managed according to the protocol (according to investigator's decision).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Vigneault, Study Chair — CHUQ - Hotel Dieu de Quebec, Quebec QC; Douglas Loblaw, Study Chair — Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto On
Locations (9):
- Canada (9):
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec

REFERENCES:
- [Result] Vigneault E, Morton G, Parulekar WR, Niazi TM, Springer CW, Barkati M, Chung P, Koll W, Kamran A, Monreal M, Ding K, Loblaw A. Randomised Phase II Feasibility Trial of Image-guided External Beam Radiotherapy With or Without High Dose Rate Brachytherapy Boost in Men with Intermediate-risk Prostate Cancer (CCTG PR15/ NCT01982786). Clin Oncol (R Coll Radiol). 2018 Sep;30(9):527-533. doi: 10.1016/j.clon.2018.05.007. Epub 2018 Jun 11. PMID 29903505

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2: IGRT 37.5 Gy in 15 fractions
  + HDR brachytherapy boost 15 Gy
  Image guided external beam radiotherapy with or without brachytherapy boost: image guided external beam radiotherapy (IGRT) or IGRT with high dose rate (HDR) brachytherapy boost
  Brachytherapy: Brachytherapy boost
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Customized [Count of Participants; unit: Participants]
  <= 65 years | 13 | 11 | 24
  > 65 years | 16 | 17 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 28 | 57
Prostate Carcinoma Disease clinical T Stage [Count of Participants; unit: Participants] — Prostate Carcinoma Disease clinical T Stage, higher stage reprent worse disease
  Participants
    T1c | 18 | 13 | 31
    T2a | 7 | 11 | 18
    T2b | 3 | 3 | 6
    T2c | 1 | 1 | 2
PSA [Count of Participants; unit: Participants]
  < 10 | 20 | 24 | 44
  10-20 | 9 | 4 | 13
The AUA Symptom Index Score [Count of Participants; unit: Participants] — The AUA Symptom Index Score, measures the bothersome the urinary symptoms. Higher value indicates of worse symptom.
  Participants
    AUA score from 0 to 9 | 18 | 21 | 39
    AUA score from 10 to 19 | 11 | 7 | 18
combined Gleason Score [Count of Participants; unit: Participants] — label the severity and stage of the prostate cancer, with higher value, the worse of the disease
  Participants
    Gleason Score of 7 | 29 | 28 | 57
    Others | 0 | 0 | 0
The ECOG Scale of Performance Status [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status, 0 indicates Fully active, while 5 means dead.
  Participants
    0 | 29 | 27 | 56
    Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Ability to Accrue Patients
Description: The ability to accrue 60 patients over an 18 month period to a study that randomizes men with intermediate-risk prostate cancer to curative intent treatment with image guided external beam radiotherapy (IGRT) or IGRT with high dose rate (HDR) brachytherapy boost within a Canadian multicentre setting.
Time Frame: 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 29 | 28
Participants | 29 | 28

2. Secondary Outcome: Number of Participants Reported Adverse Events
Description: Acute genitourinary (GU) and gastrointestinal (GI) adverse events.
Time Frame: 21 months
Population: As treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 29 | 26
Participants
  GASTROINTESTINAL DISORDERS | 1 | 0
  RENAL AND URINARY DISORDERS | 0 | 2

3. Secondary Outcome: Treatment Compliance
Description: Treatment compliance will be monitored on an ongoing basis by Central Office and the designated radiotherapy quality assurance reviewer and will be described for both arms.
Time Frame: 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 29 | 26
Participants
  Minor Deviation | 14 | 18
  Major Deviation | 3 | 2

4. Secondary Outcome: Radiotherapy Quality Assurance -Timing
Description: The time from the the time from IGRT Real Time Review Signed to IGRT Real Time Review Uploaded.
Time Frame: 5 months
Population: As treated population.
Measure: Median (Full Range); unit: Day
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 29 | 26
Day | 4 [0 to 12] | 3 [0 to 21]

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 1/29 | 2/26
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/26
Other Adverse Events (participants affected / at risk) | 0/29 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=29) | Arm 2 (N=26)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Limited follow up time, delayed side effect might not be captured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No